CLINICAL TRIAL: NCT03249064
Title: Response to Tregs in Innate Immunity Receptor LRP1 (CD91) and Tregs in Periferic Blood Mononuclear Cells in Patients With Non-segmentary Vitiligo
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-VIT-2015-69
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: VITILIGO
Keywords: TREGS; CD91; LRP1
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Periferic blood /serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitiligo untreated patients
  Interventions: Diagnostic Test: CD 91 levels; Diagnostic Test: Tregs
- Control. Patients without vitiligo
  Interventions: Diagnostic Test: CD 91 levels; Diagnostic Test: Tregs

INTERVENTIONS:
Diagnostic Test: CD 91 levels
Diagnostic Test: Tregs

SUMMARY:
This study aims to evaluate some differences in the immune system between patients with vitiligo and patients without the disease.

These differences will be evaluated by the extraction of peripheral blood that will be analyzed before the treatment and after the treatment that, in the habitual way and at the discretion of the responsible dermatologist.

Patients agreeing to participate in the study will be subjected to extraction of two tubes (20 ml) of peripheral blood (baseline) and after 12 weeks (+/- 5 days) of treatment.

Therefore, neither treatment nor follow-up visits will be modified by participation, but will be the same whether or not participate in the study.

In the case of controls, two peripheral blood tubes (20ml) will be removed in a single participation.

Patients with vitiligo will also be asked to complete questionnaires to measure stress, depression and perception of disease (PSS-10, Skindex-29, HADS, Likert) before and after 12 weeks (+/- 5 days) of therapeutic intervention .

This study will include 20 patients with active non-segmental vitiligo and 10 controls without the disease. The duration of participation in this study will be 12 weeks (+/- 5 days) for patients with vitiligo and a single participation (extraction of 20 ml of peripheral venous blood) for the controls.

ELIGIBILITY:
Inclusion Criteria:

- Patient with vitiligo without treatment

Exclusion Criteria:

* Patient with inmunosupressive disease
* Patient receiving vitiligo treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18 to 65 years-old both sex
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-09-13 (Actual)

PRIMARY OUTCOMES:
Tregs levels | Baseline
Tregs levels | 16 weeks

SECONDARY OUTCOMES:
LRP1 (CD91) levels | Baseline
LRP1 (CD91) levels | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Piquero-Casals J, Martinez-Martinez L, Alomar A, Rozas-Munoz E, Juarez C, Puig L. LRP1/CD91 is highly expressed in monocytes from patients with vitiligo - even after repigmentation. Exp Dermatol. 2021 Mar;30(3):390-395. doi: 10.1111/exd.14249. Epub 2020 Dec 14. PMID 33249636